CLINICAL TRIAL: NCT02004093
Title: A Randomized, Open-label Study of the Effect of Omnitarg in Combination With Carboplatin-based Chemotherapy Versus Carboplatin-based Therapy Alone on Treatment Response in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: A Study to Evaluate the Effect of the Combination of Pertuzumab With Carboplatin-Based Standard Chemotherapy in Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO17931
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pertuzumab; Paclitaxel; Gemcitabine; Carboplatin

ARMS (2):
- Chemotherapy + Pertuzumab (Experimental)
  Interventions: Drug: pertuzumab; Drug: paclitaxel; Drug: gemcitabine; Drug: carboplatin
- Chemotherapy (Active Comparator)
  Interventions: Drug: paclitaxel; Drug: gemcitabine; Drug: carboplatin

INTERVENTIONS:
Drug: pertuzumab — Loading dose of 840 mg IV, followed by 420 mg IV every 3 weeks
  Arms: Chemotherapy + Pertuzumab
Drug: paclitaxel — 175 mg/m2 IV every 3 weeks for 6 cycles
Drug: gemcitabine — 1000 mg/m2 IV Day 1 and 8 of each cycle for 6 cycles
Drug: carboplatin — Target AUC of 5 following paclitaxel or AUC of 4 following gemcitabine IV every 3 weeks for 6 cycles

SUMMARY:
This study will evaluate the efficacy and safety of pertuzumab in combination with carboplatin-based standard chemotherapy in patients with platinum-sensitive recurrent ovarian cancer. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed ovarian, primary peritoneal, or fallopian tube cancer;
* only 1 previous regimen, which must be platinum-based;
* platinum-sensitive disease which is defined by a progression-free interval of greater than 6 months after completion of platinum-based chemotherapy.

Exclusion Criteria:

* previous radiotherapy;
* previous treatment with an anti-cancer vaccine or any targeted therapy;
* major surgery or traumatic injury within 4 weeks of study;
* history or evidence of central nervous system metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (27):
- Belgium (3):
  - Brussels
  - Leuven
  - Wilrijk
- Canada (3):
  - Calgary, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
- Hungary (3):
  - Budapest
  - Debrecen
  - Győr
- Italy (2):
  - Parma, Emilia-Romagna
  - Milan, Lombardy
- Amsterdam, Netherlands
- Poland (2):
  - Poznan
  - Warsaw
- Russia (4):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Tomsk
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia
- United Kingdom (6):
  - Birmingham
  - London
  - Manchester
  - Plymouth
  - Sutton
  - Yeovil

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy + Pertuzumab: Participants received pertuzumab for a total of seventeen 3-week cycles and chemotherapy for a total of six 3-week cycles.
  Pertuzumab: Participants received pertuzumab 840 milligrams (mg) intravenously (IV) on Day 1 of cycle 1 and 420 mg IV on Day 1 of cycles 2 to 17; Chemotherapy consisted of EITHER:1) paclitaxel 175 mg/square meters (m^2) IV on Day 1 and carboplatin target area under the curve (AUC) 5, IV, on Day 1 followed by 2 weeks off OR 2) gemcitabine 1000 mg/m^2, IV, on Days 1 and 8 (with carboplatin target AUC of 4, IV on Day 1 only) followed by 1 week off.
- Chemotherapy: Participants received chemotherapy with EITHER: 1) paclitaxel 175 mg/m^2 on Day 1 and carboplatin AUC 5, IV, on Day 1 followed by 2 weeks off OR 2) gemcitabine 1000 mg/m^2, IV, on Days 1 and 8 (with carboplatin target AUC of 4, IV on Day 1 only) followed by 1 week off.
Period: Overall Study
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Started | 75 (Includes 1 participant who was randomized to chemotherapy group but received pertuzumab+chemotherapy) | 74
Completed | 1 | 1
Not Completed | 74 | 73
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 66 | 62
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received randomized treatment (All Treated Population, for Efficacy Analyses); 1 participant was randomized to the chemotherapy arm but received pertuzumab+chemotherapy and is thus included in this arm for all analyses.
Groups:
- Chemotherapy + Pertuzumab: Participants received pertuzumab for a total of seventeen 3-week cycles and chemotherapy for a total of six 3-week cycles.
  Pertuzumab: Participants received pertuzumab 840 mg IV on Day 1 of cycle 1 and 420 mg IV on Day 1 of cycles 2 to 17; Chemotherapy consisted of EITHER: 1) paclitaxel 175 mg/m^2 IV on Day 1 and carboplatin target AUC 5, IV, on Day 1 followed by 2 weeks off OR 2) gemcitabine 1000 mg/m^2, IV, on Days 1 and 8 (with carboplatin target AUC of 4, IV on Day 1 only) followed by 1 week off.
- Total: Total of all reporting groups
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.16) | 55.3 (11.41) | 56.7 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 149
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression was assessed according to RECIST (Response Evaluation Criteria In Solid Tumors), for participants with measurable disease, or by changes in CA 125 (Cancer Antigen 125) according to GCIG (Gynecologic Cancer Inter Group) for all participants. Participants who did not progress or died while being followed were censored at the time of the last valid tumor assessment or valid CA 125 assessment.
Time Frame: Screening and Day 15 of Cycles 2, 4, 6, and Day 15 of all cycles from Cycle 7 to 17 until disease progression up to 104 weeks
Population: All treated participants who received Randomized Treatment (All Treated Population, for Efficacy Analyses) were included in analysis.
Measure: Number; unit: percentage of participants
Groups:
- Chemotherapy + Pertuzumab: Participants received pertuzumab for a total of seventeen 3-week cycles and chemotherapy for a total of six 3-week cycles.
  Pertuzumab: Participants received pertuzumab 840 mg IV on Day 1 of cycle 1 and 420 mg IV on Day 1 of cycles 2 to 17; Chemotherapy consisted of EITHER:1) paclitaxel 175 mg/m^2 IV on Day 1 and carboplatin target AUC 5, IV, on Day 1 followed by 2 weeks off OR 2) gemcitabine 1000 mg/m^2, IV, on Days 1 and 8 (with carboplatin target AUC of 4, IV on Day 1 only) followed by 1 week off.
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
percentage of participants | 87.8 | 80.0

2. Primary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the time from first administration of study drug (Study Day 1) to documented disease progression or death, whichever occurred earlier. Disease progression was assessed according to RECIST, for participants with measurable disease, or by changes in CA 125 according to GCIG for all participants. Participants who did not progress or died while being followed were censored at the time of the last valid tumor assessment or valid CA 125 assessment.
Time Frame: as for outcome 1
Population: All treated patients who received Randomized Treatment (All Treated Population, for Efficacy Analyses) were included in analysis.
Measure: Median (Full Range); unit: weeks
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
weeks | 34.1 [31 to 38] | 40.0 [33 to 43]
Statistical Analysis 1: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.3967, Log Rank
Statistical Analysis 2: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.4552, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.3972, Wald test — p-value resulting from Wald test of null hypothesis that the hazard ratio equals (=) 1; Hazard Ratio (HR) = 1.17, 80% CI 2-sided [0.92 to 1.49]

3. Secondary Outcome: Percentage of Participants With a Best Overall Confirmed Response Based on Combined CA 125 and RECIST Measurements
Description: Response by tumor measurement occurred if there was documented and confirmed complete response (CR) or partial response (PR). For all participants, response was assessed by both the RECIST and by CA 125 levels, according to whether the participant had measurable or non-measurable disease at baseline. Response according to CA 125 levels was defined as at least a 50% reduction from baseline. The decrease had to be confirmed and maintained for at least 28 days. The confirmatory sample must have been less than or equal to the previous sample (within an assay variability of 10%). For overall response, the response categories were "response", "stable disease" and "progressive disease". Stable disease included 1) stable disease as defined by RECIST for solid tumors and 2) CA 125 levels that had not met the definition of "response" or "progressive disease".
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
percentage of participants | 74.3 | 68.0
Statistical Analysis 1: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.3943, Chi-squared; Difference in Response Rates = 6.32, 80% CI 2-sided [-3.9 to 16.6]
Statistical Analysis 2: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; Odds Ratio (OR) = 1.36, 80% CI 2-sided [0.86 to 2.17] — approximate 80% confidence interval (CI) for difference of two rates using Hauck-Anderson method

4. Secondary Outcome: Duration of Response
Description: For participants who achieved a response, the duration of response was defined as the interval between initial documentation of response to the first documentation of disease progression or death. Participants who responded and did not progress or die while on study or while being followed were censored at the last valid tumor or CA 125 measurement.
Time Frame: Day 15 of Cycles 2, 4, 6, and Day 15 of all Cycles from Cycle 7 to 17 until disease progression up to 104 weeks
Population: Only participants with a response were included in the analysis; 8 participants and 13 participants were censored in the chemotherapy + pertuzumab and chemotherapy only treatment groups, respectively.
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Chemotherapy + Pertuzumab: Participants received pertuzumab for a total of seventeen 3-week cycles and chemotherapy for a total of six 3-week cycles.Pertuzumab: Participants received pertuzumab 840 mg IV on Day 1 of cycle 1 and 420 mg IV on Day 1 of cycles 2 to 17; Chemotherapy consisted of EITHER:1) paclitaxel 175 mg/m^2 IV on Day 1 and carboplatin target AUC 5, IV, on Day 1 followed by 2 weeks off OR 2) gemcitabine 1000 mg/m^2, IV, on Days 1 and 8 (with carboplatin target AUC of 4, IV on Day 1 only) followed by 1 week off
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 47 | 38
weeks | 28.7 [22 to 48] | 37.0 [25 to 43]
Statistical Analysis 1: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.3655, Log Rank
Statistical Analysis 2: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.1319, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.3679, Wald test; p-value resulting from Wald test of null hypothesis that the hazard ratio=1; Hazard Ratio (HR) = 1.22, 80% CI 2-sided [0.92 to 1.61]

5. Secondary Outcome: Kaplan-Meier Probability of Maintaining a Response to at Least 1 Year
Time Frame: 1 year
Population: All treated patients who received Randomized Treatment (All Treated Population, for Efficacy Analyses) were included in analysis. 7 and 5 participants in the chemotherapy + pertuzumab and chemotherapy treatment groups, respectively, remained at risk.
Measure: Number; unit: percent
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 55 | 51
percent | 18 | 18

6. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was assessed according to RECIST, for participants with measurable disease, or by changes in CA 125 according to GCIG for all participants. Participants who did not progress while being followed were censored at the time of the last valid tumor assessment or valid CA 125 assessment.
Time Frame: Screening and Day 15 of Cycles 2, 4, 6, and Day 15 of all cycles from Cycle 7 to 17 until disease progression
Population: All treated participants were included in analysis
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
percentage of participants | 83.8 | 76.0

7. Secondary Outcome: Time to Progressive Disease
Description: The time to progressive disease is the interval of time from date of first dose of study medication to date of first documentation of progressive disease by either RECIST or CA 125 criteria. Participants who never progressed while being followed were censored at the last valid tumor measurement or CA 125 measurement.
Time Frame: Screening and Day 15 of Cycles 2, 4, 6, and Day 15 of all cycles from Cycle 7 to 17 until disease progression
Population: All treated patients with an event (disease progression) were included in analysis
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 62 | 57
weeks | 34.3 [27 to 48] | 37.3 [29 to 47]
Statistical Analysis 1: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.8129, Log Rank
Statistical Analysis 2: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.6920, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.8137, Wald test; p-value resulting from Wald test of null hypothesis that the hazard ratio=1; Hazard Ratio (HR) = 1.04, 80% CI 2-sided [0.82 to 1.32]

8. Secondary Outcome: Kaplan-Meier Probability of Being Progression Free at 1 Year
Time Frame: 1 year
Population: All treated patients who received Randomized Treatment (All Treated Population, for Efficacy Analyses) were included in analysis. 16 and 10 participants in the chemotherapy + pertuzumab and chemotherapy treatment groups, respectively, remained at risk.
Measure: Number; unit: percent
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 62 | 57
percent | 24 | 19

9. Primary Outcome: Kaplan-Meier Probability of No Disease or Progression at 1 Year
Description: The probability of being event free (no disease progression or death events) at 1 year in participants remaining at risk.
Time Frame: 1 year
Population: All treated patients who received Randomized Treatment (All Treated Population, for Efficacy Analyses) were included in analysis. 17 and 12 participants in the chemotherapy + pertuzumab and chemotherapy treatment groups, respectively, remained at risk.
Measure: Number; unit: percent
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
percent | 24 | 21

10. Secondary Outcome: Time To Response
Description: Time to response was the date of first dose of study medication to the date of the first documentation of response, according to CA 125 criteria for all participants or response according to RECIST criteria for participants with measurable disease. If response was evaluable by both criteria, then the date of response was for the earlier of the two events.
Time Frame: Screening and Day 15 of Cycles 2, 4, 6, and Day 15 of all cycles from Cycle 7 to 17 until 2 years after last dose of treatment
Population: Only participants with a response were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Chemotherapy + Pertuzumab: Participants received pertuzumab for a total of seventeen17 3-week cycles and chemotherapy for a total of six 3-week cycles.
  Pertuzumab: Participants received pertuzumab 840 mg IV on Day 1 of cycle 1 and 420 mg IV on Day 1 of cycles 2 to 17; Chemotherapy consisted of EITHER:1) paclitaxel 175 mg/m^2 IV on Day 1 and carboplatin target AUC 5, IV, on Day 1 followed by 2 weeks off OR 2) gemcitabine 1000 mg/m^2, IV, on Days 1 and 8 (with carboplatin target AUC of 4, IV on Day 1 only) followed by 1 week off.
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 55 | 51
weeks | 6.0 [5 to 17] | 6.3 [5 to 15]
Statistical Analysis 1: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.5726, Log Rank
Statistical Analysis 2: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.3903, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.5870, Wald test; p-value resulting from Wald test of null hypothesis that the hazard ratio=1; Hazard Ratio (HR) = 1.11, 80% CI 2-sided [0.87 to 1.43]

11. Secondary Outcome: Percentage of Participants Who Died
Time Frame: as for outcome 10
Population: All treated participants were included in analysis
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
percentage of participants | 45.9 | 41.3

12. Secondary Outcome: Overall Survival
Description: Survival was the interval of time from date of first dose of study medication to date of death at any time. Participants who had not died were censored at the date of last contact when they were known to be alive.
Time Frame: as for outcome 10
Population: All treated participants were included in analysis
Measure: Median (Full Range); unit: months
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 74 | 75
months | 28.2 [1 to 52] | NA [1 to 34] — Given the duration of follow-up at time of data analysis the median had not been reached and could not be calculated (at least 50% of patients had not died).
Statistical Analysis 1: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.9261, Log Rank
Statistical Analysis 2: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.8591, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Chemotherapy + Pertuzumab vs Chemotherapy; Test type: Superiority or Other; p = 0.9262, Wald test — p-value resulting from Wald test of null hypothesis that the hazard ratio=1; Hazard Ratio (HR) = 1.02, 80% CI 2-sided [0.74 to 1.41]

13. Secondary Outcome: Kaplan-Meier Probability of Being Alive at 1 Year
Time Frame: 1 year
Population: as for outcome 2
Measure: Number; unit: percent
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Number analyzed (Participants) | 64 | 61
percent | 88 | 85

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of randomization until 28 days after the last dose of the pertuzumab and/ or standard chemotherapy and continuously until end of study.
Groups:
- Chemotherapy + Pertuzumab: Participants received loading dose of 840mg IV Pertuzumab, followed by 420 mg IV every 3 weeks (for a total of 17 cycles), along with chemotherapy with either Paclitaxel or Gemcitabine. Paclitaxel dosage was 175 mg/m2 IV every 3 weeks for 6 cycles, followed by Carboplatin AUC of 5; Gemcitabine dosage was 1000 mg/m2 IV on day 1 and 8 of each cycle for 6 cycles followed by Carboplatin AUC of 4, IV every 3 weeks for 6 cycles.
- Chemotherapy: Participants received chemotherapy with either Paclitaxel or Gemcitabine. Paclitaxel dosage was 175 mg/m2 IV every 3 weeks for 6 cycles followed by Carboplatin AUC of 5; Gemcitabine dosage was 1000 mg/ m2 IV on day 1 and 8 of each cycle for 6 cycles followed by Carboplatin AUC of 4, IV every 3 weeks for 6 cycles.
Arm/Group | Chemotherapy + Pertuzumab | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 20/75 | 12/74
Other Adverse Events (participants affected / at risk) | 72/75 | 68/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Pertuzumab (N=75) | Chemotherapy (N=74)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Large intesting perforation (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Local swelling (General disorders) | 1 | 0
Obstruction (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Pertuzumab (N=75) | Chemotherapy (N=74)
Nausea (Gastrointestinal disorders) | 44 | 33
Diarrhoea (Gastrointestinal disorders) | 44 | 14
Vomiting (Gastrointestinal disorders) | 24 | 22
Constipation (Gastrointestinal disorders) | 20 | 22
Abdominal pain (Gastrointestinal disorders) | 18 | 14
Dyspepsia (Gastrointestinal disorders) | 9 | 6
Stomatitis (Gastrointestinal disorders) | 10 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Hemorrhoids (Gastrointestinal disorders) | 6 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 4
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 36 | 43
Anaemia (Blood and lymphatic system disorders) | 19 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 18
Leukopenia (Blood and lymphatic system disorders) | 9 | 12
Fatigue (General disorders) | 30 | 27
Asthenia (General disorders) | 9 | 10
Oedema peripheral (General disorders) | 4 | 6
Mucosal inflammation (General disorders) | 7 | 1
Pyrexia (General disorders) | 5 | 3
Chest pain (General disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 25
Rash (Skin and subcutaneous tissue disorders) | 17 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9
Nail disorder (Skin and subcutaneous tissue disorders) | 8 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 16 | 8
Dizziness (Nervous system disorders) | 9 | 6
Dysgeusia (Nervous system disorders) | 10 | 5
Neuropathy peripheral (Nervous system disorders) | 11 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 4
Paraesthesia (Nervous system disorders) | 4 | 4
Lethargy (Nervous system disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Drug hypersensitivity (Immune system disorders) | 11 | 13
Decreased appetite (Metabolism and nutrition disorders) | 19 | 4
Urinary tract infection (Infections and infestations) | 6 | 2
Cystitis (Infections and infestations) | 7 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2
Phlebitis (Vascular disorders) | 3 | 5
Flushing (Vascular disorders) | 5 | 2
Hypertension (Vascular disorders) | 6 | 0
Insomnia (Psychiatric disorders) | 6 | 5
Vaginal discharge (Reproductive system and breast disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.